CLINICAL TRIAL: NCT01583517
Title: Defining the Role of ERCP in the Evaluation and Treatment of Idiopathic Recurrent Acute Pancreatitis
Brief Title: ERCP in Idiopathic Recurrent Acute Pancreatitis
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Indiana University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Factorial | Masking: None | Purpose: Treatment
Other Study IDs: 1011003897
Record Dates: First submitted 2012-04-20; First posted 2012-04-24 (Estimated); Last update posted 2014-10-10 (Estimated); Status verified 2014-10

CONDITIONS: Recurrent Acute Pancreatitis
Keywords: Acute pancreatitis; ERCP; Sphincterotomy; Manometry; Sphincter of Oddi dysfunction
MeSH Terms: conditions — Pancreatitis; Sphincter of Oddi Dysfunction | interventions — Sphincterotomy, Endoscopic; salicylhydroxamic acid

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (4):
- Biliary sphincterotomy (Active Comparator): Cutting of the biliary sphincter muscle alone
  Interventions: Procedure: Biliary sphincterotomy
- Dual sphincterotomy (Active Comparator): Cutting of both the biliary and pancreatic sphincter muscles.
  Interventions: Procedure: Pancreatobiliary sphincterotomy
- Sham (Sham Comparator): Among patients with normal sphincter of Oddi manometry, patients will undergo no sphincterotomy (sham therapy).
  Interventions: Procedure: Sham
- Biliary sphincterotomy - Normal SOM (Active Comparator): Among patients with normal SOM, patients may be randomized to empiric biliary sphincterotomy alone.
  Interventions: Procedure: Biliary sphincterotomy

INTERVENTIONS:
Procedure: Biliary sphincterotomy — Cutting of the biliary sphincter muscle.
  Arms: Biliary sphincterotomy; Biliary sphincterotomy - Normal SOM
Procedure: Pancreatobiliary sphincterotomy — Cutting of both the biliary and pancreatic sphincter muscles.
  Arms: Dual sphincterotomy
Procedure: Sham — No sphincterotomy is performed in patients randomized to sham with normal SOM.
  Arms: Sham

SUMMARY:
The therapeutic impact of ERCP with sphincterotomy in the management of patients with idiopathic recurrent acute pancreatitis (RAP) needs further study. The investigators conducted a single center, feasibility, randomized trial to determine 1) the role of pancreatic manometry in predicting future episodes of RAP and 2) differences in the efficacy of no, biliary (BES) or pancreatobiliary (dual) endoscopic sphincterotomy (DES).

DETAILED DESCRIPTION:
Patients with idiopathic RAP, defined as ≥2 unexplained (per the treating physician) episodes of acute pancreatitis (based on standard criteria) requiring hospitalization, will be prospectively enrolled. All patients will undergo ERCP with manometry, with stratified randomization based on the assessment of pancreatic basal sphincter pressure. If <40mmHg, the patient will be randomized to sham or biliary sphincterotomy (BES). If ≥40mmHg, the patient will be randomized to BES or pancreatobiliary ("dual") sphincterotomy (DES).

Patients and physicians will not be blinded to the assignment group. Patients will be followed for up to 10 years to determine 1) incidence of RAP requiring hospitalization (using standard definitions) or 2) interval development of chronic pancreatitis (CP).

Differences between patients who did and did not develop RAP during follow-up will be compared to evaluate for factors associated with AP during follow-up.

ELIGIBILITY:
Inclusion Criteria:

* Idiopathic recurrent acute pancreatitis, defined as two or more episodes requiring hospitalization
* ERCP with SOM planned

Exclusion Criteria:

* Chronic pancreatitis
* Pancreas divisum
* Alternate etiology identified (e.g., CBD stone, IPMN)
* Inability to perform pancreatic manometry
* Pregnancy, age < 18, incarceration
* Inability to provide informed consent

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 89 (Actual)
Dates: Start 1997-09; Primary Completion 2012-04 (Actual); Study Completion 2014-10 (Actual)

PRIMARY OUTCOMES:
Recurrent acute pancreatitis | 120 months
  Patients will be followed post-ERCP for up to 10 years. The primary outcome is development of acute pancreatitis following the index ERCP, based on standard definitions.
  Acute pancreatitis is defined as new onset of pancreatic-type abdominal pain with associated elevation in serum amylase or lipase > 3 times the upper limit of normal, OR radiographic findings consistent with acute pancreatitis.

SECONDARY OUTCOMES:
Interval development of chronic pancreatitis | 120 months
  Determine the incidence of chronic pancreatitis during prolonged follow-up. Chronic pancreatitis is defined as characteristic changes on cross sectional imaging (CT or MRI/MRCP) or ERP (Cambridge classification).
Secondary assessment of risk factors for developing recurrent acute pancreatitis during follow-up | 120 months
  A post hoc analysis will be conducted to evaluate for independent factors associated with having recurrent acute pancreatitis during follow-up

CONTACTS AND LOCATIONS:
Overall Officials: Stuart Sherman, MD, Principal Investigator — Indiana University
Locations (1):
- Indiana University Health University Hospital, Indianapolis, Indiana, United States

REFERENCES:
- [Result] Cote GA, Imperiale TF, Schmidt SE, Fogel E, Lehman G, McHenry L, Watkins J, Sherman S. Similar efficacies of biliary, with or without pancreatic, sphincterotomy in treatment of idiopathic recurrent acute pancreatitis. Gastroenterology. 2012 Dec;143(6):1502-1509.e1. doi: 10.1053/j.gastro.2012.09.006. Epub 2012 Sep 11. PMID 22982183